CLINICAL TRIAL: NCT02074345
Title: A Phase III, Multicenter, Open-Label Study to Evaluate the Safety and Immunogenicity of Intramuscular TAK-816 in Healthy Infants
Brief Title: Phase III Study of Intramuscular TAK-816 in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TAK-816/OCT-002; U1111-1153-4027 (Registry Identifier: UTN); JapicCTI-142454 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteers; Haemophilus Influenzae Type b, Prevention
Keywords: Drug therapy; Safety and immunogenicity of Hib vaccine
MeSH Terms: conditions — Haemophilus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-816 0.5 mL (Experimental): Primary immunization: TAK-816 0.5 mL, intramuscular injection, once on Day 1 and every 28 days for 2 intervals (Days 29 and 57). Booster immunization: TAK-816 0.5 mL, intramuscular injection, once, 52 weeks after the third dose of primary immunization.
  Interventions: Biological: TAK-816

INTERVENTIONS:
Biological: TAK-816 — TAK-816 intramuscular injection

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of intramuscular TAK-816 in healthy Japanese infants.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called TAK-816. TAK-816 was being tested to evaluate its safety and immune response after intramuscular (IM) injection with TAK-816. This study evaluated adverse events and the seroprotection rate and geometric mean titer (GMT) of anti-polyribosylribitol phosphate (PRP)-antibodies in participants who were administered TAK-816 IM.

The study enrolled 31 participants. All participants received 3 doses of TAK-816 IM at 4-week intervals as part of the primary vaccination and 1 booster vaccination 52 weeks after the third dose of the primary vaccination.

This multi-center trial was conducted in Japan. The overall time to participate in this study was 64 weeks. Participants made multiple visits to the clinic including a final visit 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese infants.
2. Male or female infants aged 2-6 months (≥2 and <7 months) at the time of the first dose of investigational product (excluding hospitalized infants).
3. Infants whose parents or legal guardians have agreed to cooperate with the investigator during the study period.
4. The legal guardian signed and dated a written, informed consent form prior to the initiation of any study procedures.

Exclusion Criteria:

1. Any serious acute illness.
2. Any underlying cardiovascular, renal, hepatic, or hematologic disease, and/or developmental disorder.
3. History of possible Haemophilus influenzae type b (Hib) infection.
4. Previously diagnosed immunodeficiency.
5. Documented history of anaphylaxis to any ingredients of the investigational product (e.g., diphtheria toxoid).
6. A history of convulsions.
7. Previous administration of another Hib vaccine.
8. Treatment with any live vaccine during the 27 days before the first dose of TAK-816 or with any inactivated vaccine during the 6 days before dosing.
9. Prior participation in any clinical study or post-marketing clinical study.
10. Previously receipt of blood transfusions, gamma globulin preparations (except monoclonal antibody products not containing any components of Hib as antigens), systemic immunosuppressive therapy, or systemic corticosteroids, or a plan to receive any of these products during the study period.
11. Presence of thrombocytopenia or coagulopathy.
12. Children considered ineligible for the study for other reasons by the investigator or subinvestigator.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (4):
- Japan (4):
  - Kumagaya-shi, Saitama
  - Fuchu-shi, Tokyo
  - Suginami-ku, Tokyo
  - Kofu, Yamanashi

REFERENCES:
- [Derived] Togashi T, Mitsuya N, Sumino S, Takanami Y. Safety, tolerability and immunogenicity of intramuscular administration of PRP-CRM197 Hib vaccine to healthy Japanese children: An open-label trial. Vaccine. 2018 May 17;36(21):2968-2972. doi: 10.1016/j.vaccine.2018.04.040. Epub 2018 Apr 20. PMID 29685594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in Japan from 13 March 2014 to 25 March 2015.
Pre-assignment Details: Participants received open-label TAK-816 0.5 mL vaccinations, 3 initial doses and 1 booster.
Period: Overall Study
Arm/Group | TAK-816 0.5 mL
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) - all participants who received at least 1 dose of the study vaccination.
Arm/Group | TAK-816 0.5 mL
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: months] | 2.54 (0.587)
Age, Customized [Number; unit: participants]
  <2 months | 0
  ≥2 - <3 months | 22
  ≥3 - <4 months | 8
  ≥4 - <5 months | 1
  ≥5 months | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Region of Enrollment [Number; unit: participants]
  Japan | 31
Height [Mean (Standard Deviation); unit: cm] | 58.2 (2.38)
Weight [Mean (Standard Deviation); unit: kg] | 5.62 (0.551)
Anti-Polyribosylribitol Phosphate (PRP) Antibody Titer Before Primary Immunization [Number; unit: participants]
  <0.15 µg/mL | 4
  ≥0.15 µg/mL | 27
Simultaneous Vaccination of Pneumococcal Vaccine [Number; unit: participants] — Yes = pneumococcal vaccine was administered on the same day at least once in the primary immunization period.
  participants
    Yes | 0
    No | 31
Simultaneous Vaccination of Diphtheria, Tetanus, Pertussis-Inactivated Polio Vaccine (DPT-IPV) [Number; unit: participants] — Yes = DPT-IPV vaccine was administered on the same day at least once in the primary immunization period.
  participants
    Yes | 0
    No | 31
Simultaneous Vaccination of Rotavirus Vaccine [Number; unit: participants] — Yes = rotavirus vaccine was administered on the same day at least once in the primary immunization period.
  participants
    Yes | 27
    No | 4
Simultaneous Vaccination of Measles-Rubella (MR) Vaccine [Number; unit: participants] — Yes = MR vaccine was administered on the same day in the booster vaccination period.
  participants
    Yes | 0
    No | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events are defined as unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product, regardless of relationship to the medicinal product. Among these, events which are considered possibly associated with a medicinal product are defined as adverse reactions.
Time Frame: For 64 Weeks
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of the study vaccination.
Measure: Number; unit: participants
Arm/Group | TAK-816 0.5 mL
Number analyzed (Participants) | 31
participants | 31

2. Primary Outcome: Number of Participants With Adverse Reactions Related to Body Temperature (Pyrexia)
Description: Body temperature was assessed for 14 days after each vaccination and was recorded by the caregiver in a diary. Adverse reactions related body temperature was reported as pyrexia.
Time Frame: For 64 Weeks
Population: FAS included all participants who received at least 1 dose of the study vaccination.
Measure: Number; unit: participants
Arm/Group | TAK-816 0.5 mL
Number analyzed (Participants) | 31
participants | 6

3. Primary Outcome: Number of Participants With Adverse Reactions Related to Local Reactions
Description: Local Reactions were assessed 14 days after each vaccination and were recorded by the caregiver in a diary. Local reactions (injection site) were erythema, swelling, induration and pain (tenderness).
Time Frame: For 64 Weeks
Population: FAS included all participants who received at least 1 dose of the study vaccination.
Measure: Number; unit: participants
Arm/Group | TAK-816 0.5 mL
Number analyzed (Participants) | 31
participants
  Injection site erythema | 5
  Injection site swelling | 1
  Injection site induration | 1
  Injection site pain | 0

4. Primary Outcome: Number of Participants With Adverse Reactions Related to Systemic Reactions
Description: Systemic Reactions were assessed 14 days after each vaccination and were recorded by the caregiver in a diary. Systemic reactions were rash, irritability, crying, decreased appetite, vomiting, diarrhoea, somnolence (sleepiness) and insomnia (sleeplessness).
Time Frame: For 64 Weeks
Population: FAS included all participants who received at least 1 dose of the study vaccination.
Measure: Number; unit: participants
Arm/Group | TAK-816 0.5 mL
Number analyzed (Participants) | 31
participants
  Rash | 0
  Irritability | 0
  Crying | 3
  Decreased appetite | 0
  Vomiting | 1
  Diarrhoea | 5
  Somnolence | 3
  Insomnia | 2

5. Secondary Outcome: Percentage of Participant With Anti-PRP Antibody Titer ≥ 1.0 μg/mL
Description: Blood was collected and was sent to a central laboratory for the evaluation of anti-PRP antibody titer against Haemophilus influenzae type b (Hib) as an assessment of immunogenicity.
Time Frame: For 64 weeks
Population: FAS, all participants who received at least 1 dose of the study vaccination, with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-816 0.5 mL
Number analyzed (Participants) | 31
percentage of participants
  Before Primary Immunization (n=31) | 16.1 [5.452 to 33.727]
  At 4 Weeks after Primary Immunization (n=30) | 100 [88.430 to 100.000]
  Before Booster Vaccination (n=31) | 77.4 [58.904 to 90.406]
  At 4 Weeks after Booster Vaccination (n=31) | 100 [88.781 to 100.000]

6. Secondary Outcome: Percentage of Participant With Anti-PRP Antibody Titer ≥ 0.15 μg/mL
Description: Blood was collected and was sent to a central laboratory for the evaluation of anti-PRP antibody titer against Hib as an assessment of immunogenicity.
Time Frame: For 64 weeks
Population: FAS, all participants who received at least 1 dose of the study vaccination, with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-816 0.5 mL
Number analyzed (Participants) | 31
percentage of participants
  Before Primary Immunization (n=31) | 87.1 [70.166 to 96.370]
  At 4 Weeks after Primary Immunization (n=30) | 100 [88.430 to 100.000]
  Before Booster Vaccination (n=31) | 100 [88.781 to 100.000]
  At 4 Weeks after Booster Vaccination (n=31) | 100 [88.781 to 100.000]

7. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-PRP Antibody
Description: as for outcome 6
Time Frame: For 64 weeks
Population: FAS, all participants who received at least 1 dose of the study vaccination, with available data.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | TAK-816 0.5 mL
Number analyzed (Participants) | 31
μg/mL
  Before Primary Immunization (n=31) | 0.354 [0.2583 to 0.4843]
  At 4 Weeks after Primary Immunization (n=30) | 19.682 [11.3094 to 34.2544]
  Before Booster Vaccination (n=31) | 3.087 [2.0482 to 4.6518]
  At 4 Weeks after Booster Vaccination (n=31) | 51.334 [31.0689 to 84.8159]

ADVERSE EVENTS:
Time Frame: For 64 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-816 0.5 mL
Serious Adverse Events (participants affected / at risk) | 4/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-816 0.5 mL (N=31)
Inguinal hernia (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-816 0.5 mL (N=31)
Diarrhoea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 14
Injection site erythema (General disorders) | 5
Crying (General disorders) | 4
Injection site swelling (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 15
Gastroenteritis (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 3
Conjunctivitis bacterial (Infections and infestations) | 3
Exanthema subitum (Infections and infestations) | 2
Molluscum contagiosum (Infections and infestations) | 2
Somnolence (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 4
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 6
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3
Miliaria (Skin and subcutaneous tissue disorders) | 3
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.